CLINICAL TRIAL: NCT00961337
Title: Evaluation of a School-based Influenza Vaccination Program
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control, Taiwan (Other Government)
Collaborators: Public Health Bureau,Taoyan County Governmnet, Taiwan (Unknown); Education Department,Taoyan County Governmnet, Taiwan (Other)
Responsible Party: Jen-Hsiang Chuang, Centers for Disease Control, Department of Health,Taiwan, R.O.C.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DOH97-DC-2003
Record Dates: First submitted 2009-08-10; First posted 2009-08-18 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Influenza; Influenza Vaccines
Keywords: school children; influenza vaccination; vaccine effectiveness; influenza attack rate; absenteeism; Influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccination township (Experimental): Shinwu township was randomly designated as intervention township which freely vaccinated on grade 1-4 and 5-9 students.
  Interventions: Biological: Trivalent inactivated influenza vaccine
- Control townships (No Intervention): Guanyin township was designated as control township which only provide free vaccination on grade 1-4 students.

INTERVENTIONS:
Biological: Trivalent inactivated influenza vaccine — one dose
  Other Names: Brand Name: VAXIGRIP
  Arms: Vaccination township

SUMMARY:
The purpose of this study is to determine whether inactivated influenza vaccines are effective to protect school children and their households from getting influenza infection and further prevent student's absenteeism.

DETAILED DESCRIPTION:
School children were found to be the possible spreaders of the influenza. The successful prevention measure on school children was crucial for controlling the epidemic. In Taiwan, the national influenza immunization program on the grade 1-2 students started in winter, 2007. In this intervention study, the two study townships with 27 schools were included as our study population. The three time questionnaires were issued for collecting the health status of the children during the influenza season. The information on the vaccines' safety was also collected after the vaccination. The community collaborative clinics were responsible for taking the specimens.

ELIGIBILITY:
Inclusion Criteria:

* All elementary and junior high school students living in Shinwu and Guanyin townships were eligible to be enrolled into this study
* Agreed inform consent to participate in this study
* Complete three times questionaire follow-up

Exclusion Criteria:

* One junior high school in Shinwu township because it had both high school and junior high school

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7854 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Influenza attack rate | Three time points: November, December, 2008; February, 2009

SECONDARY OUTCOMES:
Children's absenteeism | before and after week 38, 2008
Vaccine effectiveness | From November, 2008 to February, 2009
Side effects after vaccination | within one week after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Hsiang Chunag, MD, MS, PhD., Principal Investigator — National Health Command Center, Centers for disease control, Department of Health, Taiwan, R.O.C
Locations (1):
- Centers for Disease Control, Taiwan, Taipei, Taiwan